CLINICAL TRIAL: NCT03901196
Title: Multi-elemental Imaging of Lung Tissues With LIBS (Laser-induced Breakdown Spectroscopy) : a Feasibility Study
Brief Title: Multi-elemental Imaging of Lung Tissues With LIBS (Laser-induced Breakdown Spectroscopy)
Acronym: MEDICO-LIBS
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC18.134; 2019-A00070-57 (Other: ID RCB)
Record Dates: First submitted 2019-03-28; First posted 2019-04-03 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Interstitial Lung Disease; Sarcoidosis; Idiopathic Pulmonary Fibrosis
Keywords: Laser Induced Breakdown Spectroscopy; Multi elemental imaging
MeSH Terms: conditions — Lung Diseases, Interstitial; Sarcoidosis; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interstitial Lung Disease: Ex : sarcoidosis, IPF
  Interventions: Diagnostic Test: Elemental analysis

INTERVENTIONS:
Diagnostic Test: Elemental analysis — LIBS multi elemental analysis of the specimen

SUMMARY:
Evaluate the feasibility of performing a multi-elemental imaging analysis of lung specimens from patients with ILDs, with an technology named LIBS (Laser Induced-Breakdown Spectroscopy)

DETAILED DESCRIPTION:
There is a major health problem due to the environmental and occupational related exposures to mineral particles, metals, and dust. The impact on health is considerable in terms of prevalence, morbidity and healthcare costs. Pathologists rarely report the presence of a possible mineral or metal-related etiology in a specimen by lack of available and convenient technology. Therefore, several respiratory diseases are considered idiopathic.

Interstitial lung disease (ILD), also known as diffuse parenchymal lung disease (DPLD) is a group of lung diseases affecting the interstitium (the tissue and space around the air sacs of the lungs). In France, 15.000 new cases of ILD are diagnosed each year. ILD may be classified according to the cause. Idiopathic ILD are ILD of unknown causes. The most frequent idiopathic ILD are sarcoidosis and idiopathic pulmonary fibrosis (IPF).These two diseases are the core topic of the present study since they may relate to important mineral or metal exposure.

The overall goal of this MEDICO-LIBS study is to evaluate the feasibility of using a laser-induced breakdown spectroscopy (LIBS)-based instrument to image(ie, identify, localize and possibly quantify) metals within selected human specimens with ILDs.

ELIGIBILITY:
Inclusion Criteria:

* Patient with ILD
* Patient informed, and agreed to participate

Exclusion Criteria:

* Patient opposed to participating in the study.
* Patient without available specimen.
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Interstitial Lung Disease
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Generation of multi-elemental images in tissues with LIBS | Within a month after reception of the biopsy by the analytical laboratory
  Evaluation of the feasibility of collecting and describing LIBS multi-elemental images of lung specimens originating from patients with ILDs

SECONDARY OUTCOMES:
Description of elemental distribution in the specimens | Within a month after reception of the biopsy by the analytical laboratory
  Comprehensive chemical characterization of both endogenous and exogenous elements for each specimen
Interpretation of the elemental maps | Within a month after reception of the biopsy by the analytical laboratory
  Understanding of the elemental distribution according to the clinical data
Comparison of the elemental distributions with results of other mineralogical investigations | Within a month after reception of the biopsy by the analytical laboratory
  Only for patients who previously benefited from other mineralogical investigations (eg, SEM-EDX), comparison of mineralogical analysis obtained with the elemental distributions obtained with LIBS

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Busser, PharmD, PhD, Principal Investigator — Grenoble Alpes University Hospital
Locations (4):
- France (4):
  - Grenoble Alpes University Hospital, Grenoble
  - CHRU de LILLE, Lille
  - CHU de Lyon HCL - GH Sud, Lyon
  - Hôpital Louis Pradel, Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Busser B, Moncayo S, Trichard F, Bonneterre V, Pinel N, Pelascini F, Dugourd P, Coll JL, D'Incan M, Charles J, Motto-Ros V, Sancey L. Characterization of foreign materials in paraffin-embedded pathological specimens using in situ multi-elemental imaging with laser spectroscopy. Mod Pathol. 2018 Mar;31(3):378-384. doi: 10.1038/modpathol.2017.152. Epub 2017 Nov 17. PMID 29148536
- [Result] Busser et al., Coord Chem Rev, 2018, 358, p70